CLINICAL TRIAL: NCT00986297
Title: Phase 1 Study of Accelerated Hypofractionated Image-Guided Radiation Therapy (IGRT) in Patients With Stage II-IV Non-Small Cell Lung Cancer and Poor Performance Status
Brief Title: Specialized Radiation Therapy in Treating Patients With Stage II, Stage III, Stage IV, or Recurrent Non-Small Cell Lung Cancer and Poor Performance Status
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000654621; SCCC-05509; 072009-061
Record Dates: First submitted 2009-09-26; First posted 2009-09-29 (Estimated); Last update posted 2020-08-20 (Actual); Status verified 2014-05

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage II non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; adenocarcinoma of the lung; adenosquamous cell lung cancer; bronchoalveolar cell lung cancer; large cell lung cancer; squamous cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung; Adenocarcinoma, Bronchiolo-Alveolar

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- arm one (Other): IGRT
  Interventions: Radiation: hypofractionated radiation therapy

INTERVENTIONS:
Radiation: hypofractionated radiation therapy — hypofractionated radiation therapy
  Other Names: IGRT

SUMMARY:
RATIONALE: Specialized radiation therapy that delivers a high dose of radiation directly to the tumor may kill more tumor cells and cause less damage to normal tissue.

PURPOSE: This phase I trial is studying the side effects and best dose of specialized radiation therapy in treating patients with stage II, stage III, stage IV, or recurrent non-small cell lung cancer and poor performance status.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To escalate the dose of accelerated hypofractionated image-guided conformal radiotherapy to a potent tumoricidal dose without exceeding the maximum-tolerated dose in patients with recurrent or stage II-IV non-small cell lung cancer and poor performance status.

Secondary

* To evaluate local regional tumor control and overall survival of patients treated with this regimen.

OUTLINE: Patients undergo accelerated hypofractionated image-guided conformal radiotherapy once daily, 5 days a week, for 3 weeks (15 fractions). Treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed up periodically for up to 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed non-small cell lung cancer

  * Stage II-IV and/or recurrent disease
  * No small cell histology
* Measurable or evaluable disease

  * Tumor not amenable to surgical resection
  * Tumor not eligible for stereotactic body radiation therapy
* No prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields

PATIENT CHARACTERISTICS:

* Zubrod performance status 2-4
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must agree to use effective contraception
* Must complete all required pretreatment evaluations

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 1 week since prior chemotherapy or chemoradiation therapy
* No concurrent chemotherapy
* No other concurrent antineoplastic therapy (including standard-fractionated radiotherapy to the chest, chemotherapy, biological therapy, vaccine therapy, and surgery) 1 week before, during, and for 1 week after completion of study therapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-10; Primary Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity | 90 days

SECONDARY OUTCOMES:
Local regional tumor control | 6 month
Overall survival | 2 year

CONTACTS AND LOCATIONS:
Overall Officials: Robert D. Timmerman, MD, Principal Investigator — Simmons Cancer Center
Locations (2):
- United States (2):
  - Stanford University, Stanford, California
  - University of Texas Southwestern Medical Center, Dallas, Texas